CLINICAL TRIAL: NCT01211626
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple Dose Study in Healthy Volunteers and Patients With Chronic Hepatitis C Viral Infection to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ANA773 Tosylate
Brief Title: Study of ANA773 in Healthy Volunteers and Patients With Hepatitis C Virus (HCV) to Assess Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ANA773-601
Record Dates: First submitted 2010-09-27; First posted 2010-09-29 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Part A, Group 1 Healthy Volunteer (Active Comparator): a single oral dose (Period 1) and multiple oral doses every other day (4 administrations) (Period 2) of 200 mg of ANA773 (n=6) or placebo (n=2)
  Interventions: Drug: ANA773; Drug: Placebo
- Part A, Group 2 Healthy Volunteer (Active Comparator): a single oral dose (Period 1) and multiple oral doses every other day (4 administrations) (Period 2) of 400 mg of ANA773 (n=6) or placebo (n=2)
  Interventions: Drug: ANA773; Drug: Placebo
- Part A, Group 3 Healthy Volunteer (Active Comparator): a single oral dose (Period 1) and multiple oral doses every other day (4 administrations) (Period 2) of 800 mg of ANA773 (n=6) or placebo (n=2)
  Interventions: Drug: ANA773; Drug: Placebo
- Part A, Group 4 Healthy Volunteer (Active Comparator): a single oral dose (Period 1) and multiple oral doses every other day (4 administrations) (Period 2) of 1200 mg of ANA773 (n=6) or placebo (n=2)
  Interventions: Drug: ANA773; Drug: Placebo
- Part A, Group 5 Healthy Volunteer (Active Comparator): a single oral dose (Period 1) and multiple oral doses every other day (4 administrations) (Period 2) of 1600 mg of ANA773 (n=6) or placebo (n=2)
  Interventions: Drug: ANA773; Drug: Placebo
- Part B, Group 6 HCV Infected Patient (Active Comparator): multiple oral doses(14 administrations) every other day of 2000 mg of ANA773 (n=6) or placebo (n=2)
  Interventions: Drug: ANA773; Drug: Placebo
- Part B, Group 7 HCV Infected Patient (Active Comparator): multiple oral doses(14 administrations) every other day of 1200 mg of ANA773 (n=6) or placebo (n=2)
  Interventions: Drug: ANA773; Drug: Placebo
- Part B, Group 8 HCV Infected Patient (Active Comparator): multiple oral doses(14 administrations) every other day of 1600 mg of ANA773 (n=6) or placebo (n=2)
  Interventions: Drug: ANA773; Drug: Placebo
- Part B, Group 9 HCV Infected Patient (Active Comparator): multiple oral doses(5 administrations) every other day of 2000 mg of ANA773 (n=8) or placebo (n=2)
  Interventions: Drug: ANA773; Drug: Placebo

INTERVENTIONS:
Drug: ANA773 — ANA773 Tosylate Capsule
Drug: Placebo — Matching Placebo Capsule

SUMMARY:
The overall study design includes two parts, Part A and Part B.

Part A evaluated ANA773 following oral administration to healthy volunteers. A total of 40 evaluable healthy volunteers were enrolled in Part A of the study.

Part B evaluated ANA773 following oral administration to patients with chronic HCV infection. A total of 34 evaluable patients were enrolled in Part B of this study in 2 study centers.

DETAILED DESCRIPTION:
Study Design:

Part A evaluated ANA773 following oral administration to healthy volunteers. A total of 40 evaluable healthy volunteers were enrolled in Part A of the study.

Part B evaluated ANA773 following oral administration to patients with chronic HCV infection. A total of 34 evaluable patients were enrolled in Part B of this study in 2 study centers.

ELIGIBILITY:
Part A Inclusion:

* Male or female, ages 18 to 65 years
* No clinically significant abnormalities
* No serious or severe chronic conditions
* Non-smokers

Part A Exclusion:

* Female subjects who are pregnant or breast-feeding
* History of significant medical condition that could interfere with study medication or associated study assessments
* History of or current drug or alcohol abuse

Part B Inclusion Criteria:

* Male or female, ages 18 to 65 years
* Diagnosed with chronic liver disease consistent with chronic hepatitis C infection for at least 6 months
* Screening HCV RNA ≥ 375,000 copies/mL or ≥ 75,000 IU/mL
* Naïve to or have relapsed from prior IFN-alpha based therapy

Part B Exclusion Criteria:

* Female subjects who are pregnant or breast-feeding
* Received anti-viral therapy or immunomodulatory therapy within 90 days prior to administration of the first dose of study medication
* Use of an investigational drug or participation in an investigational study with a licensed drug within 30 days
* History of significant medical condition that could interfere with study medication or associated study assessments
* History of or current drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and Pharmacokinetic Analysis in both Healthy Subjects and Chronic HCV Patients | Up to 41 Days
  Evaluate the Safety and Pharmacokinetic Analysis in both Healthy Subjects and Chronic HCV Patients

SECONDARY OUTCOMES:
Immunological effects in both Healthy Subjects and Chronic HCV Patients | Up to 41 days
  Evaluate the immunological effects and antiviral activity as assessed by changes in HCV RNA levels.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - PRA Clinical Research Unit, Groningen
  - Erasmus MC (EMC), Rotterdam